CLINICAL TRIAL: NCT02080338
Title: Is the 0.018-inch or the 0.022-inch Bracket Slot System More Effective in Orthodontic Treatment? A Randomized Clinical Trial.
Brief Title: 0.018 or 0.022 Bracket Slot System More Effective in Orthodontic Treatment?
Acronym: 18v22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Bearn (Other)
Collaborators: NHS Research and Development (Other Government)
Responsible Party: Sponsor-Investigator, David Bearn, Professor of Orthodontics, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20092E07; 09/S1401/56 (Registry Identifier: East of Scotland Research Ethics Service)
Record Dates: First submitted 2014-03-02; First posted 2014-03-06 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Malocclusion
Keywords: Orthodontic, Bracket slot, Effective, Randomized, Duration
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.018 bracket slot system (Experimental): Participants treated using 0.018-inch orthodontic bracket slot system
  Interventions: Device: Orthodontic bracket slot system
- 0.022 bracket slot system (Active Comparator): Participants treated using 0.022-inch orthodontic bracket slot system
  Interventions: Device: Orthodontic bracket slot system

INTERVENTIONS:
Device: Orthodontic bracket slot system — Orthodontic treatment using different orthodontic bracket slot systems

SUMMARY:
The purpose of this study is to compare the 0.018-inch and 0.022-inch bracket slot systems to determine which is more effective for orthodontic treatment .

DETAILED DESCRIPTION:
Background: Edgewise fixed orthodontic appliances are available in two different brackets slot sizes (0.018-inch and 0.022-inch). Both systems are used by clinicians worldwide with many orthodontists claiming clinical advantages and superiority of one system over the other. However, the scientific evidence supporting this area is scarce and weak. This leaves the clinician's choice of bracket slot system to be based mainly on empirical clinical preferences.

Aim: To compare the 0.018-inch and 0.022-inch conventional ligation pre-adjusted orthodontic bracket slot systems in terms of the effectiveness of treatment.

Methods/Design: Prospective, multi-centre randomised clinical trial, undertaken in the secondary care hospital environment in NHS (National Health Service) Tayside in the United Kingdom. Two hundred and sixteen orthodontic patients will be recruited in three secondary care centres in NHS Tayside, United Kingdom. The participants will be randomly allocated to treatment with either the 0.018-inch or 0.022-inch bracket slot systems (n= 108 for each group) using Victory conventional ligation pre-adjusted bracket systems (3M Unitek, Monrovia, California). Baseline records and outcome data will be collected both during and at the end of orthodontic treatment and will be assessed as follows:. Primary outcome measures: The duration of orthodontic treatment for the maxillary and mandibular arches. Secondary outcome measures: The number of scheduled appointments for the maxillary and mandibular arches, occlusal outcome (Peer Assessment Rating index), orthodontically induced inflammatory root resorption using periapical radiographs and the patient perception of wearing orthodontic appliances.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo dual arch fixed appliance orthodontic treatment in any of the three trial centers will be invited to participate in this trial by the operator planning to conduct their orthodontic treatment.

Exclusion Criteria:

* Patients who have undergone previous orthodontic treatment including fixed, removable and functional appliances.
* Patients less than 12 years old at the start of orthodontic treatment.
* Patients with orofacial clefting, severe hypodontia, and special needs patients.
* Patients undergoing orthognathic (jaw) surgery as part of their orthodontic treatment plan.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Duration of fixed appliance orthodontic treatment | Completion of orthodontic treatment, an expected average of 24 months.
  Number of months in orthodontic treatment from the start of fitting the fixed orthodontic appliance until the removal of the fixed appliance.

SECONDARY OUTCOMES:
Occlusal treatment outcome | The ooclusal outcome will be assessed at the end of orthodontic treatment, an average of 24 months.
  The quality of the treatment result will principally be measured by assessing the occlusal outcome using the Peer Assessment Rating Index (PAR Index) from study models recorded at the start and end of treatment (average 24 months).

OTHER OUTCOMES:
Biological side effect of fixed appliance orthodontic treatment | At 9 months from the start of treatment
  The amount of orthodontically induced inflammatory root resorption (OIIRR) will be investigated from periapical radiographs recorded at 9 months into active treatment.
Patient perception of wearing the fixed appliance | At six months from start of treatment
  Patient perception of wearing the fixed orthodontic appliance will be recorded using a questionnaire (Smiles Better) at 6 months from the start of treatment.
Patient perception of the of fixed appliance treatment outcome | Following the end of orthodontic treatment , an average of 24 months.
  Patient perception of the of fixed appliance treatment outcome, by comparing patient questionnaire pre-treatment and after treatment (average of 24 months).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M El-Angbawi, PhD, Principal Investigator — University of Dundee; David R Bearn, Prof, Study Chair — University of Dundee
Locations (3):
- United Kingdom (3):
  - Springfield Medical Center, Arbroath
  - Dundee Dental Hospital, Dundee
  - Perth Royal Infirmary, Perth

REFERENCES:
- [Derived] Yassir YA, El-Angbawi AM, McIntyre GT, Revie GF, Bearn DR. A randomized clinical trial of the effectiveness of 0.018-inch and 0.022-inch slot orthodontic bracket systems: part 2-quality of treatment. Eur J Orthod. 2019 Mar 29;41(2):143-153. doi: 10.1093/ejo/cjy038. PMID 30007333
- [Derived] El-Angbawi AM, Yassir YA, McIntyre GT, Revie GF, Bearn DR. A randomized clinical trial of the effectiveness of 0.018-inch and 0.022-inch slot orthodontic bracket systems: part 3-biological side-effects of treatment. Eur J Orthod. 2019 Mar 29;41(2):154-164. doi: 10.1093/ejo/cjy039. PMID 30007330
- [Derived] Yassir YA, El-Angbawi AM, McIntyre GT, Revie GF, Bearn DR. A randomized clinical trial of the effectiveness of 0.018-inch and 0.022-inch slot orthodontic bracket systems: part 1-duration of treatment. Eur J Orthod. 2019 Mar 29;41(2):133-142. doi: 10.1093/ejo/cjy037. PMID 30007300
- [Derived] El-Angbawi AM, Bearn DR, McIntyre GT. Comparing the effectiveness of the 0.018-inch versus the 0.022-inch bracket slot system in orthodontic treatment: study protocol for a randomized controlled trial. Trials. 2014 Oct 6;15:389. doi: 10.1186/1745-6215-15-389. PMID 25288125